CLINICAL TRIAL: NCT00563680
Title: A Phase 2 Study of AMG 479 in Relapsed or Refractory Ewing's Family Tumor and Desmoplastic Small Round Cell Tumors
Brief Title: QUILT-3.025: A Phase 2 Study of AMG 479 in Relapsed or Refractory Ewing's Family Tumor and Desmoplastic Small Round Cell Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NantCell, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20060283; QUILT-3.025 (Other: NantCell, Inc.)
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Askin's Tumors; Desmoplastic Small Round Cell Tumors; Estraosseous Ewing's Tumor; Ewing's Family Tumor; Ewing's Sarcoma; Primitive Neuroectodermal Tumors (PNETs); Sarcoma
Keywords: AMG 479; IGF-1R; Insulin-like growth factor; Insulin-like growth factor receptor; Ewing's; Sarcoma
MeSH Terms: conditions — Askin Tumor; Sarcoma, Ewing; Neuroectodermal Tumors, Primitive; Sarcoma; Insulin-Like Growth Factor I, Resistance To | interventions — ganitumab

ARMS (2):
- Exploratory Cohort (Experimental): If a total of two or more responses (partial and complete) in EFTs/DSRCTs are documented in this or the ongoing phase 1 study (20050118), then the study will allow enrollment of up to 10 additional EFT/DSRCT subjects who have been exposed to prior anti-IGF-1R targeting therapy.
  Interventions: Drug: AMG 479
- Main Cohort (Experimental): Subjects with relapsed Ewing's Family Tumors (EFTs) and Desmoplastic Small Round Cell Tumors (DSRCTs) who have not received prior anti-IGF-1R therapy will receive AMG 479 at 12mg/kg.
  Interventions: Drug: AMG 479

INTERVENTIONS:
Drug: AMG 479 — AMG 479 is a fully human monoclonal antibody (IgG1) against the insulin-like growth factor receptor-1 (IGF-1R). IGF-1R signaling has been shown to play a critical role in the survival of cancer cells. AMG 479 inhibits the binding of both IGF-1 and IGF-2 to IGF-1R, thus inhibiting ligand-dependent receptor activation. Inhibition of IGF-1R signaling with AMG 479 provides a potential mechanism for inhibiting tumor growth and survival.

SUMMARY:
Single-arm, open-label study of AMG 479 in up to 35 subjects with Ewing's Family Tumors (EFTs) and Desmoplastic Small Round Cell Tumors (DSRCTs) who have progressed or recurred after at least one prior chemotherapy regimen. An exploratory cohort of an additional up to 10 subjects with prior exposure to anti-IGF-1R therapy and who have progressed or recurred after at least one prior chemotherapy regimen will also be assessed.

ELIGIBILITY:
Male and female subjects ≥ 16 years of age with a diagnosis of EFT or DSRCT who have relapsed or progressed after at least one prior chemotherapeutic regimen will be eligible for this study.

Before any study-specific procedure, the appropriate written informed consent must be obtained.

Inclusion Criteria:

Disease Related Subjects with pathological or histological diagnosis of Ewing's Family Tumor or Desmoplastic Small Round Cell Tumor.

* Measurable disease as defined by RECIST.
* Documented failure of at least one prior chemotherapy regimen for their disease.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.

Demographic

* Males or females ≥ 16 years old.
* Signed written informed consent.
* Able to comply with visits and procedures.

Laboratory

* Willing to provide existing and/or newly acquired tumor samples.
* Diabetic Subjects (Type 1 or 2) must have HgbA1c < 8.0% and fasting blood glucose level < 160 mg/dL.

General

* Must be willing and able to use birth control (double barrier protection or abstinence) during and for 6 months after the study
* Prior exposure to another anti-IGF-1R therapy will only be allowed for a limited number of additional subjects (up to 10) in an exploratory cohort

Exclusion Criteria

Disease Related

* Known brain metastasis.
* History of bleeding diathesis.
* History of another malignancy.
* History of chronic hepatitis.
* Documented prior history of human immunodeficiency virus.

Laboratory

* Absolute neutrophil count < 1.5 x109/L.
* Platelet count < 100 x 109/L.
* Hemoglobin < 9 g/dL.
* PT > 1.5 x institutional upper limit of normal (IULN) or PTT > 1.0 x IULN.
* Serum creatinine > 1.5 x IULN.
* Aspartate aminotransferase (AST) > 2.5 x IULN or Alanine aminotransferase (ALT) > 2.5 x IULN (> 5.0 x if liver metastases present).
* Total bilirubin > 1.5 IULN (> 3.0 x with documented Gilbert's Syndrome)

Medication

* Antitumor treatment within 21 days of Study Day 1.
* Anticoagulation therapy within 28 days of Study Day 1.
* Major surgery within 28 days of Study Day 1.

General

* Other investigational procedures are excluded.
* Inability to tolerate intravenous administration.
* Subject is pregnant (eg, positive HCG test) or is breast feeding.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2007-10; Primary Completion 2009-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Objective response rate (Partial Response [PR] or Complete Response [CR]) as determined by RECIST | From screening to disease progression

SECONDARY OUTCOMES:
Assess the safety and tolerability of AMG 479 | From informed consent to the End of Study/Safety Follow-Up Visit
Assess the duration of response | From screening to disease progression
Assess the clinical benefit rate | From screening to disease progression
Assess the progression free survival and overall survival | From screening to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Tap WD, Demetri G, Barnette P, Desai J, Kavan P, Tozer R, Benedetto PW, Friberg G, Deng H, McCaffery I, Leitch I, Badola S, Chang S, Zhu M, Tolcher A. Phase II study of ganitumab, a fully human anti-type-1 insulin-like growth factor receptor antibody, in patients with metastatic Ewing family tumors or desmoplastic small round cell tumors. J Clin Oncol. 2012 May 20;30(15):1849-56. doi: 10.1200/JCO.2011.37.2359. Epub 2012 Apr 16. PMID 22508822
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com